CLINICAL TRIAL: NCT05970796
Title: The Feasibility and Effects of a Telehealth-delivered Physical Therapy Program for Postmenopausal Women with Urinary Incontinence
Brief Title: A Telehealth-delivered Physical Therapy Program for Postmenopausal Women with Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University (Other)
Responsible Party: Principal Investigator, Kuan-Yin Lin, Assistant Professor, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSTC 112-2314-B-002-315-
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telehealth group (Experimental): The telehealth group will receive eight sessions of individualized pelvic floor muscle training provided by a physical therapist via telehealth in 12 weeks.
  Interventions: Behavioral: Pelvic floor muscle training
- Face-to-face group (Active Comparator): The face-to-face group will be supervised by a female physical therapist who will provide pelvic floor muscle training twice a week for 12 weeks.
  Interventions: Behavioral: Pelvic floor muscle training

INTERVENTIONS:
Behavioral: Pelvic floor muscle training — The pelvic floor muscle training program will be provided via an intra-vaginal biofeedback device - Smart Kegel Trainer, which will be connected to the product application installed on the mobile phone or tablet so the participants can monitor their pelvic floor contractions in real time and directly in the application. Participants will be asked to complete three sets of 8 to 12 maximal pelvic floor muscle contractions and three to ten fast contractions per training session. The home program will be tailored to each participant and include "pelvic floor safe" exercises recommended by the Continence Foundation of Australia.

SUMMARY:
Postmenopausal women frequently report physical (hot flushes, night sweat, insomnia, vaginal dryness, sexual dysfunction, urinary incontinence, reduced fitness level, osteoporotic symptoms, sarcopenia, decreased fat free mass, etc.) and psychological (depression, anxiety, cognitive decline, etc.) symptoms. Among these symptoms, urinary incontinence is one of the most common manifestations of pelvic floor dysfunction and may significantly impact on women's quality of life. Urinary incontinence is highly prevalent (30%) in postmenopausal women and is primarily attributed to the decreased level of estrogen. Other potential risk factors for urinary incontinence after menopause include age, parity, genetic factors, pregnancy, overweight/obesity, low physical activity levels, diabetes, urinary tract infection, etc. International guidelines recommend lifestyle and behavioral change, pelvic floor muscle training and bladder training as first-line treatments for urinary incontinence in postmenopausal women. During the COVID-19 pandemic, access to and utilization of healthcare services is reduced. As travel distance has been reported as one of the strong barriers to healthcare among patients with incontinence, research has been conducted to investigate the applications and effects of telehealth. While telehealth rehabilitation may improve urinary incontinence symptoms, the field is still emerging and more studies are needed to elucidate how physical therapists can perform telehealth pelvic floor muscle training for urinary incontinence.

The objectives of this three-year study are:

1. to investigate the feasibility of a telehealth-delivered physical therapy program for postmenopausal women with urinary incontinence
2. to explore the effects of a telehealth-delivered physical therapy program on urinary incontinence symptoms, pelvic floor muscle function and quality of life in postmenopausal women with urinary incontinence
3. to compare the effectiveness of telehealth physical therapy program with face-to-face physical therapy in this population
4. to compare body composition, physical activity levels, functional capacity, grip strength, urinary incontinence symptoms, and pelvic floor muscles function in women at early versus late stage of post-menopause
5. to evaluate the relationships between duration after menopause and body composition, physical activity levels, functional capacity, grip strength, urinary incontinence symptoms, and pelvic floor muscles function

DETAILED DESCRIPTION:
This is a non-inferiority randomized controlled trial with a nested cross-sectional study and a nested qualitative interview study. Sixty community-dwelling postmenopausal women with urinary incontinence, aged >40 years, will be recruited and randomly allocated to two groups, telehealth group or face-to-face group. All groups will receive a 12-week pelvic floor muscle training. The face-to-face group will be supervised by a female physical therapist who will provide pelvic floor muscle training twice a week. The training will be adjusted according to the performance of the participant. The telehealth group will receive eight sessions of individualized pelvic floor muscle training provided by a physical therapist via telehealth in addition to a weekly telephone coaching. The baseline, post-intervention, and 3-month follow-up assessments will include feasibility outcomes, measurements of anthropometry, body composition (body composition monitor), hand grip strength (dynamometer), functional exercise capacity (six minute walk test), and pelvic floor muscle function (vaginal manometry, transperineal ultrasound and digital palpation) and two questionnaires about symptom severity of urinary incontinence and physical activity levels. This study will provide evidence of effectiveness of different delivery modes of physical therapy program for postmenopausal women with urinary incontinence and health-care professionals working with this population in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. women aged over 40 years
2. postmenopausal women: amenorrhea for longer than 12 months
3. having symptomatic UI (defined as having the Questionnaire for Urinary Incontinence Diagnosis score > 0 point)
4. being able to answer the questionnaire correctly (no language barrier or cognitive problems)
5. having no other physical or psychological problem that would interfere participation in the study
6. having access to a mobile video conference device with internet access

Exclusion Criteria:

1. women aged over 85 years old
2. receiving hormone therapy
3. having neurological conditions, malignancy for pelvic organ, overflow incontinence or voiding dysfunction
4. had received radical surgery for pelvis, sling or prolapse surgery

Ages: 40 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Number of participants consented to participate | absolute values at baseline
  Consent rate: number of participants enrolled will be divided by number of eligible patients approached
Number of intervention sessions attended | absolute values at 12 weeks
  Attendance rate: number of sessions attended will be divided by the total number of expected sessions within each treatment arm
Number of participants who remain in the study 3 months after baseline assessment | absolute values at 3 months
  Retention rate: number of participants who remain in the study at 3-month follow-up as a proportion of the total number of participants recruited at the baseline assessment
Number of participants who withdrew from the trial | absolute values at 12 weeks and 3 months
  Withdrawal rate: number of participants who withdraw from the trial after consenting divided by the number of participants who initially consent to the trial
Number of completed training sessions in relation to the scheduled sessions | absolute values at 12 weeks
  Adherence rate: the total number of exercise sessions completed as a proportion of that prescribed each week from baseline to 12 week.
Number of participants with intervention-related adverse events as assessed by CTCAE v4.0 | absolute values at 12 weeks
  Adverse events: the number of adverse or serious adverse events throughout the 12-week intervention period. Participants will be asked about any symptoms (such as pain, bleeding or itching) at each training session.
Satisfaction scale | absolute values at 12 weeks
  Satisfaction will be was assessed using a five-point Likert-scale ranging from '1 = very dissatisfied' to '5 = very satisfied'.
Acceptability scale | absolute values at 12 weeks
  Acceptability will be was assessed using a five-point Likert-scale ranging from '1 = very dissatisfied' to '5 = very satisfied'.

SECONDARY OUTCOMES:
Weight | absolute values at 12 weeks and 3 months
  Weight in kilograms will be measured using a Full Body Sensor Body Composition Monitor.
Height | absolute values at 12 weeks and 3 months
  Height in meters will be measured using a measuring tape.
Body mass index | absolute values at 12 weeks and 3 months
  Weight and height will be combined to report body mass index in kg/m^2
Body fat percentage | absolute values at 12 weeks and 3 months
  Body fat percentage will be measured using a Full Body Sensor Body Composition Monitor. Body fat percentage will be classified as 5.0 to 19.9% (low), 20.0 to 29.9% (normal), 30.0 to 34.9% (high), and 35.0% and above (very high).
Visceral fat level | absolute values at 12 weeks and 3 months
  Visceral fat level will be measured using a Full Body Sensor Body Composition Monitor. Visceral fat level will be classified as 1 to 9 (normal), 10 to 14 (high), and 15 to 30 (very high).
Skeletal muscle percentage | absolute values at 12 weeks and 3 months
  Skeletal muscle percentage will be measured using a Full Body Sensor Body Composition Monitor. Skeletal muscle percentage will be classified as 5.0 to 25.8% (low), 25.9 to 37.9% (normal), 28.0 to 29.0% (high), and 29.1 to 60.0% (very high).
Handgrip strength | absolute values at 12 weeks and 3 months
  The grip strength of dominant hand will be measured in kilograms using a Jamar Plus+ Dynamometer.
Functional exercise capacity | absolute values at 12 weeks and 3 months
  Functional exercise capacity will be assessed using six-minute walk test. The distance covered over a time of 6 minutes will be recorded in meters.
Pelvic floor muscle strength | absolute values at 12 weeks and 3 months
  Pelvic floor muscle strength will be measured using digital palpation. The results will be recorded using the modified Oxford Grading scale, which quantifies pelvic floor muscle strength as: 0, no contraction; 1, flicker; 2, weak; 3, moderate; 4, good; and 5, strong.
Bladder neck descent | absolute values at 12 weeks and 3 months
  Bladder neck descent will be measured in centimeters using a transperineal ultrasound at rest and during maximal voluntary contraction.
Anteroposterior diameter of the urogenital levator hiatus | absolute values at 12 weeks and 3 months
  Anteroposterior diameter of the urogenital levator hiatus will be measured in centimeters using a transperineal ultrasound at rest and during maximal voluntary contraction.
Anorectal angle | absolute values at 12 weeks and 3 months
  Anorectal angle will be measured using a transperineal ultrasound. The anorectal angle between the anal canal longitudinal axis and the posterior rectal line will be measured in degrees at rest and during maximal voluntary contraction.
Severity of urinary incontinence | absolute values at 12 weeks and 3 months
  The severity of urinary incontinence will be measured using the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form. The total score ranges from 0-21 with a higher score indicating greater severity of symptoms.
Physical activity levels | absolute values at 12 weeks and 3 months
  The International Physical Activity Questionnaire - Short Form will be used to measure total physical activity levels in MET minutes a week with a higher score corresponding to a higher physical activity level.

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Yin Lin, Ph.D., Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University, Taipei, Taipei, Taiwan

REFERENCES:
- [Derived] Lin KY, Chen CY, Wu PC, Huang MH, Ou YC, Kao YL, Lin KH. The feasibility and effects of a telehealth-delivered physical therapy program for postmenopausal women with urinary incontinence: A pilot mixed-methods study. Maturitas. 2025 Jun;197:108376. doi: 10.1016/j.maturitas.2025.108376. Epub 2025 Apr 23. PMID 40286562
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322